CLINICAL TRIAL: NCT06557876
Title: The Effect of Pulse Field Ablation on Atrial Mechanics Assessed by MRI and on Patient-related Outcomes in Catheter Ablation of Paroxysmal Atrial Fibrillation
Brief Title: The Effect of Pulse Field Ablation on Atrial Mechanics in Catheter Ablation of Paroxysmal Atrial Fibrillation
Acronym: PF-MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP230296
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation Paroxysmal
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: * Interventional, single center, prospective, comparative, randomized (ratio of 1:1), open-label study.
  * With 2 compared groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary vein isolation by pulse field ablation (Active Comparator)
  Interventions: Procedure: Pulmonary vein isolation by pulse field ablation
- Pulmonary vein isolation by cryoablation (Active Comparator)
  Interventions: Procedure: Pulmonary vein isolation by cryoablation

INTERVENTIONS:
Procedure: Pulmonary vein isolation by pulse field ablation — Pulse Field Ablation (PFA) is a non-thermal energy based on high voltage, ultra-short energy pulses applied selectively to cardiomyocytes.
  Arms: Pulmonary vein isolation by pulse field ablation
Procedure: Pulmonary vein isolation by cryoablation — Cryoablation is a conventional thermal energy, also delivered with a single-shot cryoballoon device.
  Arms: Pulmonary vein isolation by cryoablation

SUMMARY:
The goal of this clinical trial is to compare the effect of pulmonary vein isolation on atrial function between pulse-field and cryoablation in patients over the age of 18 with paroxysmal atrial fibrillation. The main question it aims to answer is:

• Is catheter ablation energy (pulse field ablation) revealing a better preservation of the atrial function architecture than with conventional catheter ablation technologies ?

Participants will performed 2 IRMs with injection and completed Quality of Life Questionnaires. They participate in the study for 4 months.

Researchers will compare 2 arms:

* Pulse-Field Ablation
* Cryoablation

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18
* Established diagnosis of paroxysmal fibrillation, with a I/IIa/IIb indication for catheter ablation (ESC 2020 guidelines)
* Episode of AF documented by ECG within the last 12 months
* Patient able to give written informed consent
* If female of childbearing potential, have a negative serum pregnancy test and using effective contraception
* Be affiliated with a French social security system or entitled

Exclusion Criteria:

* Non-paroxysmal atrial fibrillation
* Contraindication to oral anticoagulation
* Intracardiac thrombus
* Previous ablation in the left atrium
* Previous heart surgery
* Significant valvular heart disease defined as any moderate (grade 3) or severe (grade 4) mitral regurgitation, mitral stenosis, aortic regurgitation, aortic stenosis, tricuspid regurgitation, or tricuspid stenosis
* Contraindication to perform MRI or using the DOTAREM™ contrast product (pacemaker, defibrillator, foreign body or prosthesis, old generation heart valves, old generation ferromagnetic vascular surgical clips, percutaneous devices for endocranial aneurysms, neurosimulator, cochlear implants, automated injection device such as insulin pump, and more generally any non-removable electronic device, severe kidney disease with GFR < 30 mL/min, documented hypersensitivity to gadoteric acid or to excipients, severe claustrophobia)
* Patient on AME (state medical aid)
* Pregnant or breast-feeding female
* Patient protected by law (guardianship, tutelage measure, deprived of liberty)
* Participation in another interventional study or being in the exclusion period at the end of a previous study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-09-09 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Difference between baseline (pre-ablation) and post-ablation in the amount of left atrial fibrosis such as quantified by 3D late gadolinium enhancement (g, %) (related to primary objective) (MRI measurement) | 3 months

SECONDARY OUTCOMES:
Difference between baseline (pre-ablation) and post-ablation in global left atrial strain (%) (related to secondary objective 1) (MRI measurement) | 3 months
Difference between baseline (pre-ablation) and post-ablation in regional left atrial strains (%) (related to secondary objective 1) (MRI measurement) | 3 months
Difference between baseline (pre-ablation) and post-ablation LA adipose tissue, measured by CT (cm2, mm3, %) (related to secondary objective 1 and 2) (CT measurement) | 3 months
Difference between baseline (pre-ablation) and post-ablation left atrial flow assessed by 4D-flow MRI (related to secondary objective 3) (MRI measurement) | 3 months
Difference between baseline (pre-ablation) and post-ablation left atrial flow assessed by vortices number (related to secondary objective 3) (MRI measurement) | 3 months
Difference between baseline (pre-ablation) and post-ablation left atrial flow assessed by characterization (n) (related to secondary objective 3) (MRI measurement) | 3 months
Difference between baseline (pre-ablation) and post-ablation left atrial flow assessed by duration (ms) (related to secondary objective 3) (MRI measurement) | 3 months
Difference between baseline (pre-ablation) and post-ablation left atrial flow assessed by LA stasis (related to secondary objective 3) (MRI measurement) | 3 months
Heart rate measured the day after ablation and 3 months after (related to secondary objective 4) | 3 months
SF-36 (Short-Form-36) Physical Health Composite questionnaires measured before ablation (related to secondary objective 4). The minimum value is 0 and the maximum is 800; a higher score means a better result. | 0 day
SF-36 (Short-Form-36) Physical Health Composite questionnaires measured 15 days after ablation (related to secondary objective 4). The minimum value is 0 and the maximum is 800; a higher score means a better result. | 15 days
Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) questionnaires measured before ablation (related to secondary objective 4). The minimum value is 0 and the maximum is 100; a higher score means a better result. | 0 day
Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) questionnaires measured 15 days after ablation (related to secondary objective 4). The minimum value is 0 and the maximum is 100; a higher score means a better result. | 15 days
Numeric rating pain scale (NRS) (0-10) measured 24 hours after ablation (related to secondary objective 4) | 1 day
Numeric rating pain scale (NRS) (0-10) measured 15 days after ablation (related to secondary objective 4) | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Marine CAMUS, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Dr Mikael Laredo, Paris, France, France

IPD SHARING:
Plan to Share IPD: Undecided